CLINICAL TRIAL: NCT00149591
Title: Early and Long-Term Outcome of Elective Stenting of the Infarct-Related Artery in Patients With Viability in the Infarct-Area Early After Acute Myocardial Infarction. The VIAMI-Trial.
Brief Title: The Viability-Guided Angioplasty After Acute Myocardial Infarction-Trial (The VIAMI-Trial)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Netherlands Heart Foundation (Other)
Collaborators: The Interuniversity Cardiology Institute of the Netherlands (Other Government); Eli Lilly and Company (Industry); Boehringer Ingelheim (Industry); Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2000B026; H4S-UT-O017
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2008-09-05 (Estimated); Status verified 2006-09

CONDITIONS: Myocardial Infarction; Coronary Artery Disease
Keywords: Myocardial infarction; Viability; Coronary angioplasty; Prevention; Prognosis
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease | interventions — Angioplasty, Balloon; Stents

INTERVENTIONS:
Procedure: coronary balloon-angioplasty with stenting

SUMMARY:
The VIAMI-trial investigates the effects of balloon angioplasty with stenting of the infarct-vessel in the early phase after acute myocardial infarction. The study concerns patients who have residual viable tissue in the infarct-area after being treated with thrombolysis. It is postulated that only patients with remaining viable tissue are at high-risk for recurrent infarction or anginal attacks and that stenting of the infarct-vessel will reduce this risk considerably.

DETAILED DESCRIPTION:
Earlier studies have shown that routine angioplasty of the infarct-related coronary artery soon after thrombolysis for acute myocardial infarction did not result in a clinical benefit. This finding emphasizes the importance to select a subgroup of patients with a recent myocardial infarction, who will really benefit from angioplasty of the infarct-related artery.

Several studies have demonstrated that the presence of viability in the infarct-area early after acute myocardial infarction imposes an increased risk of new cardiac events like recurrent infarction, angina pectoris and need for coronary interventions. Therefore, it is postulated that only patients with viability in the infarct-area will benefit from angioplasty early after acute myocardial infarction.

In the VIAMI-trial patients who are admitted to the hospital with an acute myocardial infarction and who did not undergo immediate coronary angioplasty, will undergo viability testing by dobutamine-echocardiography within 3 days of admission. Patients with unequivocal signs of viability in the infarct-area will then be randomized to an invasive or a conservative treatment strategy. In the invasive strategy patients will undergo coronary angiography with the intention to perform balloon angioplasty with stenting of the infarct-related coronary artery, with concomitant use of the intravenous platelet inhibitor abciximab. In the conservative group patients will undergo coronary angiography and angioplasty only when new impending infarction or recurrent ischemia is present. In the invasive group balloon angioplasty will be performed as soon as possible after randomization. Patients without viability will not be randomized,but will participate as a control group.

ELIGIBILITY:
Inclusion Criteria:

* Admission within 6 hours of pain onset and EKG with ≥ 1 mm ST-segment elevation in two or more standard leads or ≥ 2 mm ST-elevation in two contiguous chest leads, indicative for transmural ischemia, with or without the development of new Q-waves, with myocardial necrosis proven by enzyme rise (total CPK ≥ 2x the upper normal limit).
* Patient history compatible with subacute myocardial infarction ( ≥ 6 hours), with at least signs of myocardial necrosis on the EKG (Q-waves) and a significantly increased serum level of cardiac-specific enzymes.
* Age between 18 and 80 years.
* Viability testing performed prior to coronary angiography.
* No clinical indication for an invasive procedure to be performed before viability testing

Exclusion Criteria:

* No informed consent obtained
* Unreliable follow-up
* Viability testing technically not possible
* Contra-indications for dobutamine echocardiography (heart failure, arrhythmia)
* Contra-indications for coronary angiography, such as severe diabetic nephropathy or know contrast-allergy
* Known hypersensitivity for abciximab
* Serious, life-threatening non-cardiac illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2001-04; Study Completion 2007-01

PRIMARY OUTCOMES:
Death
Recurrent myocardial infarction
Unstable angina for which hospital admission required
Analysis at 30 days, 6 months and 1 year

SECONDARY OUTCOMES:
Left ventricular function (Echocardiography)
Incidence of heart failure (NYHA)
Angina pectoris class (CCS)
Need for revascularization procedures
Analysis at 3 and 6 months and after 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gerrit Veen, MD, PhD, Principal Investigator — VU University medical center, Amsterdam, The Netherlands; Cees A Visser, MD, PhD, Study Chair — VU University medical center, Amsterdam, The Netherlands; Frans C Visser, MD, PhD, Study Director — Amsterdam UMC, location VUmc
Locations (12):
- Netherlands (12):
  - Medical Center Alkmaar (MCA), Alkmaar
  - Sint LucasAndreas Hospital, Amsterdam
  - VU University medical center, Amsterdam
  - Catharina Hospital, Eindhoven
  - Kennemer Gasthuis, Haarlem
  - Atrium Medical Center Heerlen, Heerlen
  - Hospital Hilversum, Hilversum
  - Rijnland Hospital, Leiderdorp
  - University Medical Center St. Radboud, Nijmegen
  - Waterland Hospital, Purmerend
  - Diakonessenhuis, Utrecht
  - Zaans Medical Center "De Heel", Zaandam

REFERENCES:
- [Background] Gunnar RM, Passamani ER, Bourdillon PD, Pitt B, Dixon DW, Rapaport E, Fuster V, Reeves TJ, Karp RB, Russell RO Jr, et al. Guidelines for the early management of patients with acute myocardial infarction. A report of the American College of Cardiology/American Heart Association Task Force on Assessment of Diagnostic and Therapeutic Cardiovascular Procedures (Subcommittee to Develop Guidelines for the Early Management of Patients with Acute Myocardial Infarction). J Am Coll Cardiol. 1990 Aug;16(2):249-92. doi: 10.1016/0735-1097(90)90575-a. No abstract available. PMID 2197309
- [Background] Antman EM, Anbe DT, Armstrong PW, Bates ER, Green LA, Hand M, Hochman JS, Krumholz HM, Kushner FG, Lamas GA, Mullany CJ, Ornato JP, Pearle DL, Sloan MA, Smith SC Jr, Alpert JS, Anderson JL, Faxon DP, Fuster V, Gibbons RJ, Gregoratos G, Halperin JL, Hiratzka LF, Hunt SA, Jacobs AK, Ornato JP. ACC/AHA guidelines for the management of patients with ST-elevation myocardial infarction; A report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee to Revise the 1999 Guidelines for the Management of patients with acute myocardial infarction). J Am Coll Cardiol. 2004 Aug 4;44(3):E1-E211. doi: 10.1016/j.jacc.2004.07.014. No abstract available. PMID 15358047
- [Background] Keeley EC, Boura JA, Grines CL. Primary angioplasty versus intravenous thrombolytic therapy for acute myocardial infarction: a quantitative review of 23 randomised trials. Lancet. 2003 Jan 4;361(9351):13-20. doi: 10.1016/S0140-6736(03)12113-7. PMID 12517460
- [Background] Van de Werf F, Ardissino D, Betriu A, Cokkinos DV, Falk E, Fox KA, Julian D, Lengyel M, Neumann FJ, Ruzyllo W, Thygesen C, Underwood SR, Vahanian A, Verheugt FW, Wijns W; Task Force on the Management of Acute Myocardial Infarction of the European Society of Cardiology. Management of acute myocardial infarction in patients presenting with ST-segment elevation. The Task Force on the Management of Acute Myocardial Infarction of the European Society of Cardiology. Eur Heart J. 2003 Jan;24(1):28-66. doi: 10.1016/s0195-668x(02)00618-8. No abstract available. PMID 12559937
- [Background] Hasdai D, Behar S, Wallentin L, Danchin N, Gitt AK, Boersma E, Fioretti PM, Simoons ML, Battler A. A prospective survey of the characteristics, treatments and outcomes of patients with acute coronary syndromes in Europe and the Mediterranean basin; the Euro Heart Survey of Acute Coronary Syndromes (Euro Heart Survey ACS). Eur Heart J. 2002 Aug;23(15):1190-201. doi: 10.1053/euhj.2002.3193. PMID 12127921
- [Background] Morrow DA, Antman EM, Parsons L, de Lemos JA, Cannon CP, Giugliano RP, McCabe CH, Barron HV, Braunwald E. Application of the TIMI risk score for ST-elevation MI in the National Registry of Myocardial Infarction 3. JAMA. 2001 Sep 19;286(11):1356-9. doi: 10.1001/jama.286.11.1356. PMID 11560541
- [Background] GISSI-2: a factorial randomised trial of alteplase versus streptokinase and heparin versus no heparin among 12,490 patients with acute myocardial infarction. Gruppo Italiano per lo Studio della Sopravvivenza nell'Infarto Miocardico. Lancet. 1990 Jul 14;336(8707):65-71. PMID 1975321
- [Background] ISIS-3: a randomised comparison of streptokinase vs tissue plasminogen activator vs anistreplase and of aspirin plus heparin vs aspirin alone among 41,299 cases of suspected acute myocardial infarction. ISIS-3 (Third International Study of Infarct Survival) Collaborative Group. Lancet. 1992 Mar 28;339(8796):753-70. PMID 1347801
- [Background] GUSTO Angiographic Investigators. The effects of tissue plasminogen activator, streptokinase, or both on coronary-artery patency, ventricular function, and survival after acute myocardial infarction. N Engl J Med. 1993 Nov 25;329(22):1615-22. doi: 10.1056/NEJM199311253292204. PMID 8232430
- [Background] Meijer A, Verheugt FW, Werter CJ, Lie KI, van der Pol JM, van Eenige MJ. Aspirin versus coumadin in the prevention of reocclusion and recurrent ischemia after successful thrombolysis: a prospective placebo-controlled angiographic study. Results of the APRICOT Study. Circulation. 1993 May;87(5):1524-30. doi: 10.1161/01.cir.87.5.1524. PMID 8491007
- [Background] Veen G, Meyer A, Verheugt FW, Werter CJ, de Swart H, Lie KI, van der Pol JM, Michels HR, van Eenige MJ. Culprit lesion morphology and stenosis severity in the prediction of reocclusion after coronary thrombolysis: angiographic results of the APRICOT study. Antithrombotics in the Prevention of Reocclusion in Coronary Thrombolysis. J Am Coll Cardiol. 1993 Dec;22(7):1755-62. doi: 10.1016/0735-1097(93)90754-o. PMID 8245325
- [Background] Meijer A, Verheugt FW, van Eenige MJ, Werter CJ. Left ventricular function at 3 months after successful thrombolysis. Impact of reocclusion without reinfarction on ejection fraction, regional function, and remodeling. Circulation. 1994 Oct;90(4):1706-14. doi: 10.1161/01.cir.90.4.1706. PMID 7923654
- [Background] Nijland F, Kamp O, Verheugt FW, Veen G, Visser CA. Long-term implications of reocclusion on left ventricular size and function after successful thrombolysis for first anterior myocardial infarction. Circulation. 1997 Jan 7;95(1):111-7. doi: 10.1161/01.cir.95.1.111. PMID 8994425
- [Background] TIMI Study Group. Comparison of invasive and conservative strategies after treatment with intravenous tissue plasminogen activator in acute myocardial infarction. Results of the thrombolysis in myocardial infarction (TIMI) phase II trial. N Engl J Med. 1989 Mar 9;320(10):618-27. doi: 10.1056/NEJM198903093201002. PMID 2563896
- [Background] SWIFT trial of delayed elective intervention v conservative treatment after thrombolysis with anistreplase in acute myocardial infarction. SWIFT (Should We Intervene Following Thrombolysis?) Trial Study Group. BMJ. 1991 Mar 9;302(6776):555-60. doi: 10.1136/bmj.302.6776.555. PMID 2021717
- [Background] Erbel R, Pop T, Henrichs KJ, von Olshausen K, Schuster CJ, Rupprecht HJ, Steuernagel C, Meyer J. Percutaneous transluminal coronary angioplasty after thrombolytic therapy: a prospective controlled randomized trial. J Am Coll Cardiol. 1986 Sep;8(3):485-95. doi: 10.1016/s0735-1097(86)80172-3. PMID 2943780
- [Background] Guerci AD, Gerstenblith G, Brinker JA, Chandra NC, Gottlieb SO, Bahr RD, Weiss JL, Shapiro EP, Flaherty JT, Bush DE, et al. A randomized trial of intravenous tissue plasminogen activator for acute myocardial infarction with subsequent randomization to elective coronary angioplasty. N Engl J Med. 1987 Dec 24;317(26):1613-8. doi: 10.1056/NEJM198712243172601. PMID 2960897
- [Background] Rogers WJ, Baim DS, Gore JM, Brown BG, Roberts R, Williams DO, Chesebro JH, Babb JD, Sheehan FH, Wackers FJ, et al. Comparison of immediate invasive, delayed invasive, and conservative strategies after tissue-type plasminogen activator. Results of the Thrombolysis in Myocardial Infarction (TIMI) Phase II-A trial. Circulation. 1990 May;81(5):1457-76. doi: 10.1161/01.cir.81.5.1457. PMID 2110033
- [Background] Simoons ML, Arnold AE, Betriu A, de Bono DP, Col J, Dougherty FC, von Essen R, Lambertz H, Lubsen J, Meier B, et al. Thrombolysis with tissue plasminogen activator in acute myocardial infarction: no additional benefit from immediate percutaneous coronary angioplasty. Lancet. 1988 Jan 30;1(8579):197-203. doi: 10.1016/s0140-6736(88)91062-8. PMID 2893037
- [Background] Topol EJ, Califf RM, George BS, Kereiakes DJ, Abbottsmith CW, Candela RJ, Lee KL, Pitt B, Stack RS, O'Neill WW. A randomized trial of immediate versus delayed elective angioplasty after intravenous tissue plasminogen activator in acute myocardial infarction. N Engl J Med. 1987 Sep 3;317(10):581-8. doi: 10.1056/NEJM198709033171001. PMID 2956516
- [Background] Froelicher VF, Perdue S, Pewen W, Risch M. Application of meta-analysis using an electronic spread sheet to exercise testing in patients after myocardial infarction. Am J Med. 1987 Dec;83(6):1045-54. doi: 10.1016/0002-9343(87)90940-5. PMID 3332565
- [Background] Basu S, Senior R, Raval U, Lahiri A. Superiority of nitrate-enhanced 201Tl over conventional redistribution 201Tl imaging for prognostic evaluation after myocardial infarction and thrombolysis. Circulation. 1997 Nov 4;96(9):2932-7. doi: 10.1161/01.cir.96.9.2932. PMID 9386159
- [Background] Bigi R, Desideri A, Bax JJ, Galati A, Coletta C, Fiorentini C, Fioretti PM. Prognostic interaction between viability and residual myocardial ischemia by dobutamine stress echocardiography in patients with acute myocardial infarction and mildly impaired left ventricular function. Am J Cardiol. 2001 Feb 1;87(3):283-8. doi: 10.1016/s0002-9149(00)01359-x. PMID 11165961
- [Background] Huitink JM, Visser FC, Bax JJ, van Lingen A, Groenveld AB, Teule GJ, Visser CA. Predictive value of planar 18F-fluorodeoxyglucose imaging for cardiac events in patients after acute myocardial infarction. Am J Cardiol. 1998 May 1;81(9):1072-7. doi: 10.1016/s0002-9149(98)00143-x. PMID 9605044
- [Background] Lee KS, Marwick TH, Cook SA, Go RT, Fix JS, James KB, Sapp SK, MacIntyre WJ, Thomas JD. Prognosis of patients with left ventricular dysfunction, with and without viable myocardium after myocardial infarction. Relative efficacy of medical therapy and revascularization. Circulation. 1994 Dec;90(6):2687-94. doi: 10.1161/01.cir.90.6.2687. PMID 7994809
- [Background] Tieleman RG, Van Gelder IC, Crijns HJ, De Kam PJ, Van Den Berg MP, Haaksma J, Van Der Woude HJ, Allessie MA. Early recurrences of atrial fibrillation after electrical cardioversion: a result of fibrillation-induced electrical remodeling of the atria? J Am Coll Cardiol. 1998 Jan;31(1):167-73. doi: 10.1016/s0735-1097(97)00455-5. PMID 9426036
- [Background] Nijland F, Kamp O, Verhorst PM, de Voogt WG, Visser CA. In-hospital and long-term prognostic value of viable myocardium detected by dobutamine echocardiography early after acute myocardial infarction and its relation to indicators of left ventricular systolic dysfunction. Am J Cardiol. 2001 Nov 1;88(9):949-55. doi: 10.1016/s0002-9149(01)01968-3. PMID 11703987
- [Background] Petretta M, Cuocolo A, Bonaduce D, Nicolai E, Cardei S, Berardino S, Ianniciello A, Apicella C, Bianchi V, Salvatore M. Incremental prognostic value of thallium reinjection after stress-redistribution imaging in patients with previous myocardial infarction and left ventricular dysfunction. J Nucl Med. 1997 Feb;38(2):195-200. PMID 9025734
- [Background] Previtali M, Fetiveau R, Lanzarini L, Cavalotti C, Klersy C. Prognostic value of myocardial viability and ischemia detected by dobutamine stress echocardiography early after acute myocardial infarction treated with thrombolysis. J Am Coll Cardiol. 1998 Aug;32(2):380-6. doi: 10.1016/s0735-1097(98)00243-5. PMID 9708464
- [Background] Salustri A, Ciavatti M, Seccareccia F, Palamara A. Prediction of cardiac events after uncomplicated acute myocardial infarction by clinical variables and dobutamine stress test. J Am Coll Cardiol. 1999 Aug;34(2):435-40. doi: 10.1016/s0735-1097(99)00232-6. PMID 10440156
- [Background] Sicari R, Picano E, Landi P, Pingitore A, Bigi R, Coletta C, Heyman J, Casazza F, Previtali M, Mathias W Jr, Dodi C, Minardi G, Lowenstein J, Garyfallidis X, Cortigiani L, Morales MA, Raciti M. Prognostic value of dobutamine-atropine stress echocardiography early after acute myocardial infarction. Echo Dobutamine International Cooperative (EDIC) Study. J Am Coll Cardiol. 1997 Feb;29(2):254-60. doi: 10.1016/s0735-1097(96)00484-6. PMID 9014975
- [Background] Iskander S, Iskandrian AE. Prognostic utility of myocardial viability assessment. Am J Cardiol. 1999 Mar 1;83(5):696-702, A7. doi: 10.1016/s0002-9149(98)00973-4. PMID 10080421
- [Background] Carlos ME, Smart SC, Wynsen JC, Sagar KB. Dobutamine stress echocardiography for risk stratification after myocardial infarction. Circulation. 1997 Mar 18;95(6):1402-10. doi: 10.1161/01.cir.95.6.1402. PMID 9118506
- [Background] Picano E, Sicari R, Landi P, Cortigiani L, Bigi R, Coletta C, Galati A, Heyman J, Mattioli R, Previtali M, Mathias W Jr, Dodi C, Minardi G, Lowenstein J, Seveso G, Pingitore A, Salustri A, Raciti M. Prognostic value of myocardial viability in medically treated patients with global left ventricular dysfunction early after an acute uncomplicated myocardial infarction: a dobutamine stress echocardiographic study. Circulation. 1998 Sep 15;98(11):1078-84. doi: 10.1161/01.cir.98.11.1078. PMID 9736594
- [Background] Samad BA, Frick M, Hojer J, Urstad MJ. Early low-dose dobutamine echocardiography predicts late functional recovery after thrombolyzed acute myocardial infarction. Am Heart J. 1999 Mar;137(3):489-93. doi: 10.1016/s0002-8703(99)70497-7. PMID 10047631
- [Background] Yoshida K, Gould KL. Quantitative relation of myocardial infarct size and myocardial viability by positron emission tomography to left ventricular ejection fraction and 3-year mortality with and without revascularization. J Am Coll Cardiol. 1993 Oct;22(4):984-97. doi: 10.1016/0735-1097(93)90407-r. PMID 8409073
- [Background] Nijland F, Kamp O, Verhorst PM, de Voogt WG, Bosch HG, Visser CA. Myocardial viability: impact on left ventricular dilatation after acute myocardial infarction. Heart. 2002 Jan;87(1):17-22. doi: 10.1136/heart.87.1.17. PMID 11751656
- [Background] Bax JJ, Wijns W, Cornel JH, Visser FC, Boersma E, Fioretti PM. Accuracy of currently available techniques for prediction of functional recovery after revascularization in patients with left ventricular dysfunction due to chronic coronary artery disease: comparison of pooled data. J Am Coll Cardiol. 1997 Nov 15;30(6):1451-60. doi: 10.1016/s0735-1097(97)00352-5. PMID 9362401
- [Background] EPILOG Investigators. Platelet glycoprotein IIb/IIIa receptor blockade and low-dose heparin during percutaneous coronary revascularization. N Engl J Med. 1997 Jun 12;336(24):1689-96. doi: 10.1056/NEJM199706123362401. PMID 9182212
- [Background] EPISTENT Investigators. Randomised placebo-controlled and balloon-angioplasty-controlled trial to assess safety of coronary stenting with use of platelet glycoprotein-IIb/IIIa blockade. Lancet. 1998 Jul 11;352(9122):87-92. doi: 10.1016/s0140-6736(98)06113-3. PMID 9672272
- [Background] Montalescot G, Barragan P, Wittenberg O, Ecollan P, Elhadad S, Villain P, Boulenc JM, Morice MC, Maillard L, Pansieri M, Choussat R, Pinton P; ADMIRAL Investigators. Abciximab before Direct Angioplasty and Stenting in Myocardial Infarction Regarding Acute and Long-Term Follow-up. Platelet glycoprotein IIb/IIIa inhibition with coronary stenting for acute myocardial infarction. N Engl J Med. 2001 Jun 21;344(25):1895-903. doi: 10.1056/NEJM200106213442503. PMID 11419426
- [Background] Mehta SR, Yusuf S, Peters RJ, Bertrand ME, Lewis BS, Natarajan MK, Malmberg K, Rupprecht H, Zhao F, Chrolavicius S, Copland I, Fox KA; Clopidogrel in Unstable angina to prevent Recurrent Events trial (CURE) Investigators. Effects of pretreatment with clopidogrel and aspirin followed by long-term therapy in patients undergoing percutaneous coronary intervention: the PCI-CURE study. Lancet. 2001 Aug 18;358(9281):527-33. doi: 10.1016/s0140-6736(01)05701-4. PMID 11520521
- [Background] Steinhubl SR, Berger PB, Mann JT 3rd, Fry ET, DeLago A, Wilmer C, Topol EJ; CREDO Investigators. Clopidogrel for the Reduction of Events During Observation. Early and sustained dual oral antiplatelet therapy following percutaneous coronary intervention: a randomized controlled trial. JAMA. 2002 Nov 20;288(19):2411-20. doi: 10.1001/jama.288.19.2411. PMID 12435254
- [Background] Rao AK, Pratt C, Berke A, Jaffe A, Ockene I, Schreiber TL, Bell WR, Knatterud G, Robertson TL, Terrin ML. Thrombolysis in Myocardial Infarction (TIMI) Trial--phase I: hemorrhagic manifestations and changes in plasma fibrinogen and the fibrinolytic system in patients treated with recombinant tissue plasminogen activator and streptokinase. J Am Coll Cardiol. 1988 Jan;11(1):1-11. doi: 10.1016/0735-1097(88)90158-1. PMID 3121710
- [Background] Weissman NJ, Levangie MW, Newell JB, Guerrero JL, Weyman AE, Picard MH. Effect of beta-adrenergic receptor blockade on the physiologic response to dobutamine stress echocardiography. Am Heart J. 1995 Aug;130(2):248-53. doi: 10.1016/0002-8703(95)90436-0. PMID 7631603
- [Background] Schiller NB, Shah PM, Crawford M, DeMaria A, Devereux R, Feigenbaum H, Gutgesell H, Reichek N, Sahn D, Schnittger I, et al. Recommendations for quantitation of the left ventricle by two-dimensional echocardiography. American Society of Echocardiography Committee on Standards, Subcommittee on Quantitation of Two-Dimensional Echocardiograms. J Am Soc Echocardiogr. 1989 Sep-Oct;2(5):358-67. doi: 10.1016/s0894-7317(89)80014-8. PMID 2698218
- [Derived] van Loon RB, Veen G, Kamp O, Baur LH, van Rossum AC. Left ventricular remodeling after acute myocardial infarction: the influence of viability and revascularization - an echocardiographic substudy of the VIAMI-trial. Trials. 2014 Aug 18;15:329. doi: 10.1186/1745-6215-15-329. PMID 25135364
- [Derived] van Loon RB, Veen G, Baur LH, Kamp O, Bronzwaer JG, Twisk JW, Verheugt FW, van Rossum AC. Improved clinical outcome after invasive management of patients with recent myocardial infarction and proven myocardial viability: primary results of a randomized controlled trial (VIAMI-trial). Trials. 2012 Jan 3;13:1. doi: 10.1186/1745-6215-13-1. PMID 22214287